CLINICAL TRIAL: NCT03152500
Title: A Randomised, Subject-masked Evaluation of Stability After Implantation of Two Different Lens Models: FEMTIS-study
Brief Title: Evaluation of Stability After Implantation of Two Different Lens Models: FEMTIS-study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Oculentis (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL58195.068.16
Record Dates: First submitted 2017-05-08; First posted 2017-05-15 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2017-05

CONDITIONS: Cataract
Keywords: IOL; Stability; FEMTIS IOL; Acrysof IOL; FLACS; Capsulotomy
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FEMTIS IOL (Experimental): The FEMTIS-IOL has a special haptic system that allows the lens to clamp into the capsulorrhexis.
  Interventions: Device: FEMTIS 313G IOL
- Acrysof IOL (Active Comparator): The Acrysof IOL has a flexible haptic design that keeps the IOL stable and centered in the capsular bag
  Interventions: Device: Acrysof SN60WF IOL

INTERVENTIONS:
Device: FEMTIS 313G IOL — Haptic design that enclaves the capsulorrhexis
  Arms: FEMTIS IOL
Device: Acrysof SN60WF IOL — IOL in the bag
  Arms: Acrysof IOL

SUMMARY:
In this study the investigators will investigate the stability of lens position and the visual outcome after implantation of the new FEMTIS-IOL using FLACS capsulotomy compared to conventional placement of the IOL in the capsular bag. So far, there are no published studies using the FEMTIS-IOL. Therefore, the investigators will perform this randomized control trial.

DETAILED DESCRIPTION:
Cataract is a clouding of the crystalline lens which causes vision loss and blindness if untreated. Cataract surgery is the most frequently performed surgical intervention in medicine with an incidence of 880 surgeries per 100.000 population in 2010 amounting to a total number of over 160.000 surgeries per year in the Netherlands.1,3 The number of individuals with cataracts is predicted to reach 30 million by the year 2020.2 Due to aging of the general population this number of cataracts will only grow in the future.

For the last decade conventional phacoemulsification cataract surgery (CPCS) is the dominant form of cataract surgery in developed countries, accounting for over 90 percent of these procedures.4 The basic phacoemulsification procedure has remained largely unchanged over the past 20 years, including a series of steps: creating corneal incision, capsulorhexis and lensfragmentation.4 Although highly successful, each of the steps mentioned above are created manually which affects the safety and effectiveness of the procedure.

Since the first human eye was treated by femtosecond laser cataract surgery in 2008, the femtosecond-laser assisted cataract surgery (FLACS) became an innovative growing new technology in the world of cataract surgery.4-7 Femtosecond-lasers are capable of performing some of the most delicate and essential key steps during cataract surgery: capsulotomy, lens fragmentation, and corneal incisions. 'Automating' these steps and performing them with increased precision could lead to an improved quality of capsulotomy, easier lens fragmentation, and more precisely positioned corneal incisions, which in turn, lead to improved visual and refractive outcomes, a decrease in intra- and postoperative complication rates, and increased quality of life.

In order to remove the crystallized human lens, a circular opening in the capsular lens bag, capsulotomy, needs to be created. After removing the lens an intraocular lens (IOL) can be inserted in the empty capsule bag. However, one of the factors affecting postoperative achieved visual acuity and refraction, is the behaviour of this IOL in the capsular bag. Preoperative measurements need to be obtained in order to calculate the required IOL. One of the challenges of these IOL calculations is determining exactly where in the eye the IOL will end up, the effective lens position (ELP). The position of the IOL is crucial for the IOL's general performance because it influences the postoperative IOL tilt, decentration, and posterior capsule opacification (PCO). Considering the anatomical variety between patients, the predictability of an individual's ELP remains an educated guess.

The ELP, and therefore the amount of IOL tilt, decentration and PCO, of an IOL is mainly influenced by the interaction between the IOL and the lens capsule, especially during the time of capsule shrinkage. Theoretically, the positive optical effect of an IOL is lost when there is more than 7 degrees of tilt or more than 0.4 mm of decentration.8 Furthermore, studies have shown the effect of axial displacement of an IOL on refractive error. There is approximately 1.25 D change per millimetre of the IOL's longitudinal displacement.9 This reflects the importance of a stable and predictable ELP.

As mentioned above, the anatomy of an individual's eye is unique and therefore, each ELP will be different when placing the IOL in the capsular bag. Therefore, a new lens type has been developed: the FEMTIS® FB-313 laser lens (FEMTIS-IOL, Oculentis). This IOL has a special haptic system and is designed to be clasped in the capsular bag opening and therefore, the ELP of this IOL is theoretically more stable and predictable, resulting in a higher predictability of refractive and visual outcomes. However, in order to provide as much stability as possible a (nearly) perfect capsulotomy is needed. Several comparative studies have shown that femtosecond-lasers produce a more precise, circular, reproducible, and better centered capsulotomy compared to conventional manual capsulorhexis.6-7 The combination between the femtosecond-assisted capsulotomy and the implantation of a FEMTIS-IOL in the capsular opening, could definitely contribute to the search of perfection in cataract surgery.

In this study the investigators will investigate the stability of lens position and the visual outcome after implantation of the new FEMTIS-IOL using FLACS capsulotomy compared to conventional placement of the IOL in the capsular bag. So far, there are no published studies using the FEMTIS-IOL. Therefore, the investigators will perform this randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 40 years of age
* Cataracta Senilis
* Expected postoperative astigmatism ≤ 0.75 D (combination with FLACS AK is tolerated up to 1.25 D preoperative astigmatism)
* IOL power calculation between +10.00 D and 27.00 D
* Expected postoperative best-corrected visual acuity of logMAR +0.3 or better
* If eligible, availability to undergo second eye surgery within 2 weeks of the first eye surgery
* Willing and able to comply with scheduled visits and other study procedures
* Signed informed consent.

Exclusion Criteria:

* Traumatic cataract
* Previous corneal surgery and/or reshaping
* Clinically significant corneal endothelial dystrophy (e.g., Fuchs' dystrophy)
* Irregular astigmatism
* History of corneal disease (e.g., herpes simplex, herpes zoster keratitis, etc.)
* Extensive age related macular degeneration (atrophic or exudative age-related macular degeneration or numerous soft drusen)
* Extensive visual field loss (e.g., glaucoma, history of cerebral vascular accidents, etc.)
* Extensive diabetic macular disease
* Amblyopia, strabismus
* Keratoconus
* Pseudoexfoliation syndrome or other capsule or zonular abnormalities that could affect postoperative centration or tilt of the IOL
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils, or pupils that do not dilate at least 3.5 mm under mesopic/scotopic conditions)
* Cognitive, cerebral or concentration disorders (e.g. dementia, Parkinson, etc.)
* Suturing of incision required at time of surgery
* Complications during surgery of the first eye.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Decentration:To compare the amount of decentration between FEMTIS IOL versus a standard monofocal IOL (Acrysof monofocal IOL) using retro-illumination slitlamp photographs | 13 weeks/3months
  To compare the amount of decentration between FEMTIS IOL versus a standard monofocal IOL (Acrysof monofocal IOL) using retro-illumination slitlamp photographs

SECONDARY OUTCOMES:
Rotation stability | 13 weeks/3months
  To compare rotation stability between both IOls using retro-illumination slitlamp photographs
Tilt: To compare the amount of tilt between both IOls using Scheimpflug images | 13 weeks/3months
  To compare the amount of tilt between both IOls using Scheimpflug images
Visual outcomes | 13 weeks/3months
  Uncorrected (UDVA) and corrected (CDVA) distance visual acuity using ETDRS reading charts.

CONTACTS AND LOCATIONS:
Overall Officials: Rudy Nuijts, MD PhD, Principal Investigator — University Eye Clinic Maastricht, Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared